CLINICAL TRIAL: NCT02339532
Title: Neoadjuvant Phase II Trial Combining [3 FEC 100 Followed by 3 Docetaxel Associated With Trastuzumab Plus Pertuzumab] or [6 Docetaxel, Carboplatin Associated With Trastuzumab Plus Pertuzumab] According to TOP2A Status in Patients With T1c Operable, HER2-positive Breast Cancer
Brief Title: Neoadjuvant Phase II Trial in Patients With T1c Operable, HER2-positive Breast Cancer According to TOP2A Status
Acronym: NeoTOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEP13
Record Dates: First submitted 2014-12-14; First posted 2015-01-15 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: HER2-positive; non-metastatic; TOP2A
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Trastuzumab; pertuzumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOP2A amplified (Experimental): If TOP2A amplified: FEC x 3 then THP x 3 3 cycles of FEC 100 administered IV q3w
  * 5-Fluorouracil (5-FU) 500 mg/m²
  * Epirubicin 100 mg/m²
  * Cyclophosphamide 500 mg/m²
  Followed by 3 cycles of Trastuzumab-Pertuzumab-Docetaxel:
  * Trastuzumab 8 mg/kg loading dose administered intravenously (IV) followed by 6 mg/kg IV q3w in subsequent cycles.
  * Pertuzumab 840 mg loading dose administered IV followed by 420 mg IV q3w in subsequent cycles.
  * DOCETAXEL 75 mg/m² IV escalating at 100 mg/m² IV as tolerated q3w
  Interventions: Drug: FEC100; Drug: Docetaxel; Drug: Trastuzumab; Drug: Pertuzumab
- TOP2A not amplified (Experimental): If TOP2A not amplified: TCHP x 6 TCHP administered IV q3w for 6 cycles
  * Trastuzumab 8 mg/kg loading dose administered IV followed by 6 mg/kg IV q3w in subsequent cycles.
  * Pertuzumab 840 mg loading dose administered IV followed by 420 mg IV q3w in subsequent cycles.
  * DOCETAXEL 75 mg/m² IV q3w
  * CARBOPLATIN AUC 6 IV q3w
  The Calvert formula will be used to calculate the dose of carboplatin:
  Dose (mg) = target AUC (mg/mL x min) x [GFR mL/min + 25] Dose (mg) = 6 x [GFR mL/min + 25] NOTE: the Calvert formula gives the dose in mg, not mg/m². GFR, glomerular filtration rate The maximum dose of CARBOPLATIN must not exceed 900 mg.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Carboplatin

INTERVENTIONS:
Drug: FEC100 — 3 cycles of FEC 100 administered IV q3w
  * 5-Fluorouracil (5-FU) 500 mg/m²
  * Epirubicin 100 mg/m²
  * Cyclophosphamide 500 mg/m²
  Arms: TOP2A amplified
Drug: Docetaxel — TOP2A amplified : DOCETAXEL 75 mg/m² IV escalating at 100 mg/m² IV as tolerated q3w TOP2A not amplified : DOCETAXEL 75 mg/m² IV
Drug: Trastuzumab — Trastuzumab 8 mg/kg loading dose administered intravenously (IV) followed by 6 mg/kg IV q3w in subsequent cycles.
Drug: Pertuzumab — Pertuzumab 840 mg loading dose administered IV followed by 420 mg IV q3w in subsequent cycles.
Drug: Carboplatin — CARBOPLATIN AUC 6 IV q3w
  Arms: TOP2A not amplified

SUMMARY:
The main objective of this multicenter study will therefore be to evaluate pathologic complete response rates of an anthracycline-based regimen [FEC 100 - TAXOTERE® - HERCEPTIN® - PERTUZUMAB] and a non anthracycline-based regimen [TAXOTERE® - CARBOPLATINE - HERCEPTIN® - PERTUZUMAB] according to the presence or not of TOP2A gene amplification in a population of breast cancer patients with HER2 overexpression.

A very important objective of the study will be the evaluation of biomarkers that predict response to treatment.

DETAILED DESCRIPTION:
In this phase II study, we propose a treatment strategy that not only takes advantage of the complementary action of trastuzumab and pertuzumab but also the relevance of an anthracycline-based regimen. Indeed, besides the cardiac toxicity that can be induced by these three agents, anthracycline chemotherapy may not confer benefit to all patients.

The underlying scientific hypothesis is based on data from the NEOSPHERE neoadjuvant trial showing that addition of pertuzumab to trastuzumab plus docetaxel improved the pCR rate (46% versus 29% without pertuzumab) in T2-T3 tumors. Therefore, we hypothesize that for smaller tumors (T1c), the pCR rate should be higher, on the order of 60% in patients with the coamplification (with anthracycline therapy) and 55% for the group without coamplification (without anthracycline therapy). The sample size of 90 patients (45 per group) planned for the phase II study will allow 15% precision with the expected pCR rates of 60% (95%CI: 45%-75%) for patients with coamplification and 55% (95%CI: 40%-70%) for those without coamplification. In addition, exploratory analyses will aim to identify predictive markers of pCR in order to target biologically defined subpopulations in which pCR rates might even be higher.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18;
* Patient has histologically confirmed breast cancer, with a clinical tumour diameter of > 1 cm (cT1c, cT2-3 or T4a)-
* Any N status
* No clinically or radiologically detectable metastases (M0);
* HR negative (both ER and PR < 10% by IHC); for T1c status, otherwise HR negative or positive
* Her-2 positive (i.e. IHC score 3+ or FISH/SISH/CISH positive);
* Performance status ≤ 1 (according to WHO criteria);
* Patients not previously treated by surgery, radiotherapy, hormone therapy or chemotherapy;
* Hæmatology: Absolute neutrophil count (ANC) ≥1,500/mm³; Platelets ≥100,000/mm³; Total white blood cell count (WBC) ≥3.000/mm³; Hb> 9g/dl;
* Hepatic Function: Total bilirubin ≤1.5 time the upper normal limit (UNL); ASAT ≤ 1.5xUNL; ALAT ≤ 1.5xUNL; Alkaline phosphatase ≤ 2.5xUNL;
* Renal Function: Serum creatinine ≤1.5xUNL (and if Serum creatinine >1.5xUNL, Creatinine clearance ≥50 mL/min (MDRD formula);
* Metabolic Function: Magnesium ≥ lower limit of normal; Calcium ≥ lower limit of normal;
* Patient with not controlled heart disease and for whom anthracyclines are not contraindicated. Cardiac ejection fraction ≥50% measured by MUGA or ECHO done within 4 weeks before inclusion;
* Patient agreeing to use effective contraception during and for ≥ 7 months after completion of study treatment;
* Patient able to comply with the protocol;
* Patient must have signed a written informed consent form prior to any study specific procedures;
* Patient must be affiliated to a Social Health Insurance.

Exclusion Criteria:

* Bilateral or multifocal breast cancer;
* Non-measurable tumour;
* Any form of breast cancer other than those described in the inclusion criteria, particularly inflammatory and/or overlooked forms (T4b or T4d);
* HER2 negative status (i.e. IHC score 0 or 1+, or IHC score 2+ and FISH/SISH/CISH negative);
* RH positive (ER or PR ≥ 10% by IHC) ;
* Patient has a history of second cancer, with exception of in situ cervical cancer or basocellular skin cancer which is regarded as cured;
* Patient has already been treated for new breast cancer;
* Patients have already undergone surgery for their disease or have had primary axillary dissection;
* Prior docetaxel administration or anti-HER2 antibody therapy (e.g.: trastuzumab or pertuzumab);
* Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, such as, but not limited to:

  * Heart or kidney failure, medullary, respiratory or liver failure, dyspnea
  * Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia, poorly controlled hypertension) ≤ 1 year before enrollment
  * Uncontrolled diabetes
  * Significant neurological or psychiatric abnormalities
  * Symptomatic or progressive disorder of the central nervous system (CNS) or metastasis at the initial check-up.
  * Peripheral neuropathy > grade 2
  * Acute urinary infection, ongoing hemorrhagic cystitis;
* Patients with a known history of HIV seropositivity;
* Sensitivity to any of the study medications or any of the ingredients or excipients of these medications;
* Patients receiving of the concomitant medications with phenytoin;
* Patients who received any other investigational drugs within 30 days of initiation of treatment and/or during the study;
* Must not have had a major surgical procedure within 30 days of initiation of treatment;
* Pregnant women, women who are likely to become pregnant or are breast-feeding;
* Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Patients with history of non compliance to medical regimens or unwilling or unable to comply with the protocol;
* Individual deprived of liberty or placed under the authority of a tutor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Pathological complete response according to Chevallier classification | 20 weeks
  on surgical specimen and lymph nodes at the time of the surgery

SECONDARY OUTCOMES:
Predictive factors of response to both treatment regimens (anthracycline-based and non anthracycline-based regimens) | 20 weeks
  on surgical specimen and lymph nodes at the time of the surgery
Pathological complete response (pCR), according to Sataloff's classification | 20 weeks
  on surgical specimen and lymph nodes at the time of the surgery
Clinical and radiological response according to the WHO criteria | after two cycles of treatment and after the end of treatment
  on mammography and breast echography
Toxicity according to NCI CTC-AE v4.0 criteria | during on-treatment period (defined as the period from the first dose of study medication up to 30 days of the last dose
  according the occurrence of adverse events and toxicities assessed every week
Progression-free survival | up to 60 months
  The PFS is defined as the time from the first administration of treatment to progression or death of any cause, if progression has not been documented.
Overall survival | up to 60 months
  The OS is defined as the time from the first administration of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Ange MOURET REYNIER, Principal Investigator — Centre Jean Perrin
Locations (12):
- France (12):
  - Institut de Cancerologie de L'Ouest - Site Paul Papin, Angers
  - Centre Hospitalier Regional Universitaire de Brest - Hôpital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Chu de Grenoble - Hopital Michallon, Grenoble
  - Chu de Limoges - Hôpital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Regional Du Cancer Montpellier Val D'Aurelle, Montpellier
  - Institut de Cancerologie de L'Ouest - Site Rene Gauducheau, Saint-Herblain
  - Hopital D'Instructions Des Armees, Saint-Mandé
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancerologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Ginzac A, Molnar I, Durando X, Motte Rouge T, Petit T, D'hondt V, Campone M, Bonichon-Lamichhane N, Venat Bouvet L, Levy C, Augereau P, Pistilli B, Arsene O, Jouannaud C, Nguyen S, Cayre A, Tixier L, Mahier Ait Oukhatar C, Nabholtz JM, Penault-Llorca F, Mouret-Reynier MA. Neoadjuvant anthracycline-based (5-FEC) or anthracycline-free (docetaxel/carboplatin) chemotherapy plus trastuzumab and pertuzmab in HER2 + BC patients according to their TOP2A: a multicentre, open-label, non-randomized phase II trial. Breast Cancer Res Treat. 2024 Jun;205(2):267-279. doi: 10.1007/s10549-024-07285-y. Epub 2024 Mar 7. PMID 38453781